CLINICAL TRIAL: NCT00699101
Title: A Multi-site Prospective, Non Randomized Study Utilizing the Conture® Multi-Lumen Balloon (MLB) Breast Brachytherapy Applicator to Deliver Accelerated Partial Breast Irradiation: Analysis of Dosimetric Success, Local Tumor Control, Cosmetic Outcome, Acute and Chronic Toxicity, and Clinical Scenarios for Optimal Use
Brief Title: Using the Conture® Multi-Lumen Balloon to Deliver Accelerated Partial Breast Brachytherapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: SenoRx, Inc. (Industry)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENORX-S07-002
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Conture®; Brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Conture Multi-Lumen Balloon
  Interventions: Device: Conture Multi-Lumen Balloon

INTERVENTIONS:
Device: Conture Multi-Lumen Balloon — Placement of the balloon in a separate procedure using ultrasound guidance after surgery for breast cancer.

SUMMARY:
This multiple site, prospective, non-randomized study has been designed to compile information on the efficacy of the Contura™ MLB in delivering APBI in appropriately selected patients through evaluation of dosimetric success as compared with a single central lumen balloon device and through treatment outcomes.

DETAILED DESCRIPTION:
Data collected during this study will include baseline patient demographics, information related to the time of implant, radiation therapy details, and removal of the device as well as recurrence data, cosmetic outcomes and toxicities. The patient's follow-up data will be collected during the patient's standard follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent
* Age 50 or older at diagnosis
* Life expectancy greater than 10 years (excluding diagnosis of breast cancer).
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (negative surgical margins per NSABP criteria).
* On histologic examination, the tumor must be DCIS or invasive breast carcinoma. For patients with invasive breast cancer, an axillary staging procedure must be performed. Either:

  1. sentinel node biopsy (SNB) alone if sentinel node(s) is/are negative; or
  2. axillary dissection (minimum of six axillary nodes removed); and
  3. the axillary node(s) must be pathologically negative.
* The T stage must be Tis, T1, or T2. If T2, the tumor must be ≤ 3.0 cm in maximum diameter.
* Estrogen receptor positive tumor

Exclusion Criteria:

* Age < 50 at diagnosis (regardless of histology)
* Pregnant or breast-feeding (if appropriate, patient must use birth control during the study)
* Active collagen-vascular disease
* Paget's disease of the breast
* History of DCIS or invasive breast cancer
* Prior breast or thoracic RT for any condition
* Multicentric carcinoma (DCIS or invasive)
* Synchronous bilateral invasive or non-invasive breast cancer
* Surgical margins that cannot be microscopically assessed or that are positive or close
* Positive axillary node(s)
* T stage of T2 with the tumor > 3 cm in maximum diameter or a T stage > 3
* Estrogen receptor negative tumor

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dosimetric efficacy of the Contura™ MLB with the historical efficacy rate of a single central lumen balloon device. | 5 years

SECONDARY OUTCOMES:
Quantify the dosimetric improvement of multi-lumen use over single lumen use through dosimetric comparison. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Arthur, MD, Study Chair — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Cuttino LW, Arthur DW, Vicini F, Todor D, Julian T, Mukhopadhyay N. Long-term results from the Contura multilumen balloon breast brachytherapy catheter phase 4 registry trial. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1025-9. doi: 10.1016/j.ijrobp.2014.08.341. Epub 2014 Oct 13. PMID 25442036